CLINICAL TRIAL: NCT04241354
Title: A Comparison of Platelet-rich Plasma Treatment to the Intra-articular vs. Intra- and Extra-articular Environments in Patients Diagnosed With Hip Osteoarthritis
Brief Title: A Comparison of PRP Treatment to the IA vs. IA and EA Environments in Patients Diagnosed With Hip Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regenerative Orthopedics and Sports Medicine (Industry)
Collaborators: EmCyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSM-HO-001
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis; Degeneration
Keywords: platelet-rich plasma; leukocyte poor platelet rich plasma; PRP; hip osteoarthritis; osteoarthritis; Regenerative orthopedics and sports medicine; ROSM; EmCyte
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-articular LP-PRP Injection (Active Comparator): A single injection of leukocyte poor platelet rich plasma (LP-PRP) will be administered to the intra-articular space under ultrasound guidance at the treatment visit.
  Interventions: Biological: Leukocyte-poor platelet rich plasma
- Intra- and extra- articular LP-PRP Injection (Experimental): A single injection of LP-PRP will be administered to the intra- articular space and the extra- articular structures under ultrasound guidance at the first visit.
  Interventions: Biological: Leukocyte-poor platelet rich plasma

INTERVENTIONS:
Biological: Leukocyte-poor platelet rich plasma — Platelet rich plasma was prepared using PurePRP Supra Physiologic Protocol A preparation [EmCyte Corp. Fort Myers FL].

SUMMARY:
The purpose of this study is to evaluate the efficacy of one leukocyte-poor platelet-rich plasma (LP-PRP) injection to the intra-articular (IA) space in comparison to one LP-PRP injection to the IA space with an additional injection into the surrounding extra-articular (EA) structures for the treatment of hip OA (Kellgren Lawrence Grades 1-3). Our hypothesis is that patients receiving both IA and EA LP-PRP injections will have equivalent improvements on HOOS JR and VAS scores over a 12-month period compared to those in the active comparator group (IA LP-PRP injection).

DETAILED DESCRIPTION:
A novel comprehensive approach through which the joint and its surrounding structures are treated as an integrated system may offer a clinically superior treatment to hip osteoarthritis (OA) compared to only an intra-articular (IA) infiltration. The efficacy of autologous leukocyte-poor platelet-rich plasma (LP-PRP) for the treatment of OA is a growing area of regenerative orthopedic research.

The purpose of this study is to determine if a LP-PRP treatment to both the IA space and EA supporting capsular ligament and tendon structures provides a significant clinical benefit when compared to an IA treatment alone. In this clinical study of 84 patients, both study arms receive effective treatments that are supported by sound medical evidence, making this an ethically strong model to address our hypothesis.

This is a multi-site, randomized, comparative study of LP-PRP treatment into the IA space versus the IA space and EA hip structures. This study is sponsored by Regenerative Orthopedics and Sports Medicine (ROSM) and EmCyte Corporation. Patients who meet the study criteria with at least mild pain as indicated by >25/100 on a 100mm visual analogue scale (VAS) (Sanchez et al. 2011), or <80/100 on HOOS JR with radiographic evidence of Kellgren-Lawrence grades 1-3 hip OA will be invited to participate in this study.

The preparation of PRP is a simple tissue fractionation using centrifugation with EmCyte PurePRP Supraphysiologic SP kit [EmCyte Corp. Fort Myers FL]. Platelet quantification analysis is performed using the Horiba ABX Micros ES 60 [Plymouth Medical]. Primary outcome measures are indicated by overall hip pain severity by HOOS JR and VAS patient reported outcome measures.

ELIGIBILITY:
Inclusion:

1. Symptomatic OA of hip (K-L Grade 1-3) documented by x-ray taken within the past 6 months
2. Male or female age 30 - 65 at time of enrollment
3. Patients must have adequate immune system function with no known immunodeficiency
4. disease
5. Has not had a corticosteroid injection in the past 6 months
6. Has not used non-steroidal anti-inflammatory 7 days prior to treatment and has not used oral
7. corticosteroids 30 days prior to treatment
8. If on chronic anticoagulant medication, we will follow the recommendations of the physician
9. managing their anticoagulant medication
10. Willing and able to participate for the entire study period
11. No evidence of current systemic infection or illness (eg. fever, malaise, etc.) and no evidence
12. of skin infection in the areas where the injection will be performed

Exclusion:

1. Patients have been diagnosed with an autoimmune disease, diabetes, rheumatoid arthritis,
2. hematologic conditions predisposing to bleeding disorders or platelet dysfunction, Paget's disease of femur or ilium, avascular necrosis (AVN) of the femoral head, infectious arthritis, Lyme disease.
3. Previous reparative cellular/ orthobiologics /PRP injection
4. ≥7mm hip effusion as measured on ultrasound at the femoral neck
5. K-L Grade 4 OA x-ray documented
6. Patient has a history of alcohol or drug abuse within the six months prior to enrolment in the study
7. Patients who had intra-articular treatment with corticosteroids within 6 months of randomization in this study
8. Patient received more than 2 previous intra- or extra-articular corticosteroid injections to the affected hip.
9. Patients who are pregnant or nursing at the time of consent
10. Patients who have had anorexia, chronic insomnia, immunocompromised state, and/ or are on immunosuppressive medication
11. Neoplastic cancer within 5 years prior to screening and no evidence of recurrence, except for cutaneous (basal cell and squamous cell) cancer treated with excision
12. History of chemotherapy within the past 3 years or radiation therapy to the involved hip area
13. Patients with inflammatory arthritic conditions (e.g. rheumatoid arthritis)
14. Patients who have had previous intervention to the hip except for labral repair/ reconstruction and/ or femoral neck osteoplasty or acetabular osteoplasty without microfracture.
15. Additional disabilities in any of the lower limbs that would interfere with any of the clinical assessments.
16. Use of NSAID 7 days prior to treatment or oral or subcutaneous corticosteroids 30 days prior
17. Patients with a BMI over 35
18. Deformity or dysplasia (i.e. Legg Calve Perthes or DDH) other than FAI.
19. Patients with systemic infection, hematological conditions, malignancy, blood borne diseases, allergies to lidocaine.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-08-25 (Estimated)

PRIMARY OUTCOMES:
Hip Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | baseline
  This is a patient-reported outcome measure for which scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating optimal hip health.
Numeric Rating Scale | baseline
  This is a patient-reported outcome measure. Scores range from 0 to 10 with score of 0 indicating no pain and a score of 10 indicating most intense pain.
Numeric Rating Scale | 6 weeks
  This is a patient-reported outcome measure. Scores range from 0 to 10 with score of 0 indicating no pain and a score of 10 indicating most intense pain.
Numeric Rating Scale | 4 months
  This is a patient-reported outcome measure. Scores range from 0 to 10 with score of 0 indicating no pain and a score of 10 indicating most intense pain.
Numeric Rating Scale | 6 months
  This is a patient-reported outcome measure. Scores range from 0 to 10 with score of 0 indicating no pain and a score of 10 indicating most intense pain.
Numeric Rating Scale | 12 months
  This is a patient-reported outcome measure. Scores range from 0 to 10 with score of 0 indicating no pain and a score of 10 indicating most intense pain.
Hip Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | 6 weeks
  This is a patient-reported outcome measure for which scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating optimal hip health.
Hip Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | 4 months
  This is a patient-reported outcome measure for which scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating optimal hip health.
Hip Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | 6 months
  This is a patient-reported outcome measure for which scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating optimal hip health.
Hip Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | 12 months
  This is a patient-reported outcome measure for which scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating optimal hip health.

CONTACTS AND LOCATIONS:
Overall Officials: Sean W Mulvaney, MD, Principal Investigator — Regenerative Orthopedics and Sports Medicine
Locations (1):
- Regenerative Orthopedics and Sports Medicine, North Bethesda, Maryland, United States